CLINICAL TRIAL: NCT04333160
Title: A Multicenter, Randomized, Double-blind, Placebo- and Active-Controlled Phase III Study on the Safety and Efficacy of a Single Intra-articular Administration of JTA-004 in Symptomatic Knee Osteoarthritis
Brief Title: Phase III Study on the Safety and Efficacy of a Single Intra-articular Administration of JTA-004 in Symptomatic Knee Osteoarthritis
Acronym: JTA-KOA2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bone Therapeutics S.A (Industry)
Collaborators: Nordic Bioscience A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 000014/BT
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Symptomatic Osteoarthritis of the Knee
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- JTA-004 (Experimental): single knee intra-articular injection of JTA-004 solution (2ml)
  Interventions: Drug: JTA-004
- placebo (Placebo Comparator): single knee intra-articular injection of saline solution (2ml)
  Interventions: Other: placebo
- Hylan G-F 20 (Active Comparator): single knee intra-articular injection of Hylan G-F 20 (6ml)
  Interventions: Device: Hylan G-F 20

INTERVENTIONS:
Drug: JTA-004 — Patients will undergo a single intra-articular injection of JTA-004 into the knee joint
  Arms: JTA-004
Device: Hylan G-F 20 — Patients will undergo a single intra-articular injection of Hylan G-F 20 into the knee joint
  Arms: Hylan G-F 20
Other: placebo — Patients will undergo a single intra-articular injection of placebo into the knee joint
  Other Names: saline solution
  Arms: placebo

SUMMARY:
Osteoarthritis is a degenerative, chronic, and progressive joint disease considered as the most common joint disorder worldwide. In healthy joints, there is a continuous process of natural breakdown and repair of cartilage. This process becomes disrupted in OA, leading to degeneration and loss of articular cartilage, along with other joint changes, including subchondral bone remodeling, osteophyte formation, thickening of the capsule and sometimes inflammation of the synovia. JTA-004 is a plasma protein solution supplemented with HA and clonidine developed as a single IA injection for the treatment of knee OA. Local administration of JTA-004 into the joint cavity is intended to relieve chronic pain in subjects suffering from knee OA and discomfort associated with the IA administration.

The JTA-004 Phase III study is a placebo and active-controlled, randomized, double-blind study to evaluate the potential of a single, intra-articular injection of JTA-004 to reduce osteoarthritic pain in the knee at 3 months compared to placebo or active comparator. The study is expected to enrol 742 patients with mild to moderate symptomatic knee osteoarthritis in 22 centres in 6 European countries and Hong Kong SAR.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory (able to walk unassisted, the use of a crutch or a walking stick (only one) is allowed if already used at screening but should be avoided during the study up to the 6-month follow-up visit)
* Diagnosed with primary knee OA, fulfilling the following American College of Rheumatology (ACR) criteria at the target knee:

  * Pain present for most days of the preceding month
  * Morning stiffness < 30 minutes
  * Kellgren-Lawrence grade II or III (confirmed by appropriate X-rays taken within 6 months prior to screening visit)
* Target knee pain ≥ 200 mm and ≤ 400 mm out of 500 mm on the WOMAC® VA3.1 pain questionnaire (sum of 5 questions) at screening and baseline
* Insufficient/failed response or intolerance to analgesics and/or non-steroidal anti-inflammatory drugs (NSAIDs) as reported by the subject
* Willing and able to abstain from initiation of physical therapy and of use of knee braces at the target knee up to the 6-month follow-up visit (a subject undergoing physical therapy or using knee braces at a stable frequency for at least 2 weeks prior to screening is allowed to continue at same frequency (frequency increase is not allowed))
* Capable to understand and comply with study requirements and to provide a written, dated, and signed informed consent prior to any study procedure for participation in the study and transmission of personal "pseudo-anonymized" data

Exclusion Criteria:

1. History of trauma or surgery or arthroscopy at the target knee within 12 months before inclusion
2. Concomitant inflammatory disease or other conditions affecting the joints (e.g., infectious arthritis, rheumatoid arthritis, psoriatic arthritis or spondyloarthropathy, Paget's disease, hemochromatosis…)
3. Any target knee abnormality that could impact safety or efficacy assessment
4. Microcrystalline arthropathies: chondrocalcinosis/calcium pyrophosphate dihydrate disease (pseudo-gout) or gout if believed likely to interfere with the study endpoints, in the opinion of the Investigator
5. Clinically significant valgus/varus deformities at the Investigator's discretion
6. Any musculoskeletal condition (such as symptomatic hip OA, amputation, neurologic disorder, chronic back pain with or without radiculopathy, sciatica) that would impede measurement of efficacy at target knee
7. Contralateral knee pain equal to or exceeding the pain in the target knee (on the WOMAC® VA3.1 pain questionnaire) at screening and/or baseline
8. Knee arthroplasty planned within 12 months after the screening visit Current or previous diagnoses, signs and/or symptoms
9. Uncontrolled diabetes mellitus (hemoglobin A1c [HbA1c] > 10% or > 86 mmol/mol), end-stage hepatic or renal disease (severe and clinically significant abnormalities according to local laboratory ranges) documented in the subject's file
10. Any relevant cardiovascular disease (severe coronary insufficiency, conduction disturbances, recent myocardial infarction, cerebrovascular disease) or any clinically significant electrocardiogram (ECG) abnormality as judged by the Investigator
11. Subject with neuropathic pain or chronic pain syndrome including fibromyalgia
12. Current (or within the last 5 years prior to entering the study) history of solid or hematological neoplasia or bone marrow transplantation (except for basal cell carcinoma and completely excised squamous cell carcinoma)
13. Other severe acute or chronic medical or psychiatric conditions or pre-dispositions or laboratory abnormalities, as judged by the Investigator
14. Current or past history of coagulation disorders (according to local laboratory ranges), as judged by the Investigator
15. Hypersensitivity to any components of hyaluronic acid (HA)-based injection products
16. Hypersensitivity to human biological material including blood and blood-derived products, potential excipients and residues from manufacturing process, documented clinically or by laboratory tests
17. Hypersensitivity to avian proteins Current or previous treatment
18. Participation in another clinical trial within 3 months prior to screening (within 1 year prior to screening if disease-modifying OA drug (DMOAD) received and if the Investigator considers it could impact the safety or efficacy assessment)
19. Subject previously treated with JTA-004 within 2 years prior to screening
20. Subject treated with intra-articular viscosupplement or blood-derived product (e.g., platelet-rich plasma) injection in the target knee within 6 months prior to screening
21. Subject treated with intra-articular glucocorticoid injection in the target knee within 4 months prior to screening
22. Subject having started the use of slow acting drugs for OA such as glucosamine, glucosamine sulfate, chondroitin sulfate, diacerein, curcumin, soybean/avocado extracts or related products within 1 month prior to screening
23. Current chemo-, radio- or immuno-cancer-therapy or immunosuppressive therapy
24. Chronic (≥ 3 days/week within the last 3 months) use of opioids other than weak opioids (such as codeine, dihydrocodeine, tramadol…)
25. Chronic (> 15 consecutive days) use of systemic steroids Safety aspects concerning female subjects of childbearing potential
26. Breast-feeding
27. Pregnancy
28. Woman with positive pregnancy test
29. Woman not willing or not able to use a highly effective contraceptive method during the 6-month active follow-up period. Highly effective birth control methods are:

    1. Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
    2. Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
    3. Intrauterine device
    4. Intrauterine hormone-releasing system
    5. Bilateral tubal occlusion Other exclusion criteria
30. Body Mass Index (BMI) of 40 kg/m2 or greater at baseline
31. Signs of an active drug or alcohol dependence, serious current illness, mental illness or any other factors which may interfere with subject's ability to understand and comply with study requirements, as judged by the Investigator
32. Life expectancy less than 12 months at screenin

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 746 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
knee pain | 3 months
  Difference between JTA-004 and placebo in mean change from baseline in knee pain at Month 3 using the Western Ontario McMaster University (WOMAC®) Visual Analogue 3.1 pain subscale (subscale A; score 0 (no-pain)-100 (worst imaginable pain) mm).

SECONDARY OUTCOMES:
knee pain | 6 months
  Difference between JTA-004 and placebo in mean change from baseline in knee pain at Month 6 using the WOMAC® Visual Analogue 3.1 pain subscale (subscale A; score 0 (no-pain)-100 (worst imaginable pain) mm))
Knee pain | 3 months
  Difference between JTA-004 and active comparator in mean change from baseline in knee pain at Month 3 using the WOMAC® Visual Analogue 3.1 pain subscale (subscale A; score 0 (no-pain)-100 (worst imaginable pain) mm))
knee physical function | 3 months
  Difference between JTA-004 and placebo in mean change from baseline in knee physical function at Month 3 using the WOMAC® Visual Analogue 3.1 physical function subscale (subscale C; score 0 (no-pain)-100 (worst imaginable pain) mm))
Patient Global assessment | 3 months
  Difference between JTA-004 and placebo in mean change from baseline in Patient Global Assessment at Month 3
physical function | 6 months
  Difference between JTA-004 and placebo in mean change from baseline in knee physical function at Month 6 using the WOMAC® Visual Analogue 3.1 physical function subscale (subscale C; 0 (no-pain)-100 (worst imaginable pain) mm))
subject global health and well-being | 3 months
  Difference between JTA-004 and placebo in mean change from baseline in subject global health and well-being score at Month 3 using the EQ-5D-5L questionnaire
responder rate | 3 months
  Difference between JTA-004 and placebo in responder rate (defined as ≥ 30% pain intensity reduction) at Month 3

CONTACTS AND LOCATIONS:
Locations (22):
- Belgium (4):
  - Cliniques universitaires Saint-Luc (UCL), Brussels
  - UZ Leuven University Hospitals Leuven, Leuven
  - CHU Liège, Liège
  - CHU Ambroise Paré, Mons
- Czechia (3):
  - CCR Brno, s.r.o, Brno
  - CCR Czech, a.s, Pardubice
  - CCR Prague s.r.o, Prague
- Denmark (4):
  - The Parker Institute, Frederiksberg
  - Sanos Clinic, Gandrup
  - Sanos Clinic, Herlev
  - Sanos Clinic, Vejle
- Hong Kong Center for Clinical Research, Hong Kong, Hong Kong
- Moldova (2):
  - "Timofei Mosneaga" Republican Clinical Hospital, Sectia Reumatologie,, Chisinau
  - RTL SM SRL / Institutul de Cardiologie, sectia consultativa, Chisinau
- Poland (7):
  - PL35, Bytom
  - PL37, Gdansk
  - PL36, Katowice
  - PL31, Nadarzyn
  - PL32, Poznan
  - PL33, Poznan
  - PL34, Swidnica
- St Pancras Clinical Research, London, United Kingdom